CLINICAL TRIAL: NCT02364804
Title: A Study to Evaluate the Efficacy of Anti-emetic Drug Aprepitant Upon the Combination Chemotherapy of Nedaplatin and Docetaxel for Non-small Cell Lung Cancer
Brief Title: A Study to Evaluate the Efficacy of Anti-emetic Drug Upon the Combination Chemotherapy for Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Shiga University (Other)
Responsible Party: Principal Investigator, Yataro Daigo, Professor, Shiga University
Other Study IDs: 24-20
Record Dates: First submitted 2015-02-02; First posted 2015-02-18 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Aprepitant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aprepitant — The incidence and grade of chemotherapy-induced nausea and vomit (CINV) will be assessed in patients receiving Aprepitant for the prevention of CINV upon the combination chemotherapy of nedaplatin and docetaxel for NSCLC. These data will be compared with those surveyed retrospectively in patients who had received the combination chemotherapy with anti-emetic agents but Aprepitant.
  Other Names: Emend

SUMMARY:
The purpose of this study is to evaluate the efficacy of anti-emetic drug Aprepitant upon the combination chemotherapy of nedaplatin and docetaxel for non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of anti-emetic drug Aprepitant upon the combination chemotherapy of nedaplatin and docetaxel for non-small cell lung cancer (NSCLC). The incidence and grade of chemotherapy-induced nausea and vomit (CINV) will be assessed in patients receiving Aprepitant for the prevention of CINV upon the combination chemotherapy of nedaplatin and docetaxel for NSCLC. These data will be compared with those surveyed retrospectively in patients who had received the combination chemotherapy with anti-emetic agents except Aprepitant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receive the combination chemotherapy of nedaplatin and docetaxel as a treatment or an adjuvant therapy for non-small cell lung cancer.
2. ECOG performance status 0-1.
3. Aged 20-79 years old.
4. Laboratory values as follows 4000/mm3 < WBC < 12000/mm3, neutrophil count > 2000/mm3, platelet count > 100000/mm3, hemoglobin > 9.5g/dL, asparate transaminase < 2.5 X cutoff value, alanine transaminase < 2.5 X cutoff value, total bilirubin < 1.5g/dL, Serum creatinine < cutoff value, PaO2 > 60 Torr.
5. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Allergy against polysorbert 80 or platinum-containing drugs.
2. Severe complications (i.e. ischemic heart diseases required treatment, arrhythmia, myocardial infarction within 6 months, liver cirrhosis, uncontrolled diabetes, and hemorrhagic tendency).
3. Active and uncontrolled infectious disease.
4. Massive pleural or pericardial effusion.
5. Other malignancy requiring treatment.
6. Active interstitial pneumonitis or its past historyBreastfeeding and Pregnancy (woman of child bearing potential)
7. Peripheral nerve disorder.
8. Pregnant or lactating women.
9. Concurrent administration of pimozide.
10. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients who receive the combination chemotherapy of nedaplatin and docetaxel
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of anti-emetic drug efficacy: Incidence and grade of nausea/vomiting | Fifteen days after beginning of each cycle of chemotherapy

SECONDARY OUTCOMES:
Influence on clinical outcome: Survival | Participants will be followed for 3 years after the last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yataro Daigo, MD, PhD, Principal Investigator — Shiga University of Medical Science
Locations (1):
- Shiga University of Medical Science Hospital, Ōtsu, Shiga, Japan